CLINICAL TRIAL: NCT01314781
Title: Comparison of Solifenacin Combined With Pelvic Floor Muscle and Whole Body Vibration Training With Solifenacin Alone in Patients With Overactive Bladder Syndrome. - A Prospective Randomized Parallel Group Trial
Brief Title: Therapy of the Overactive Bladder Syndrome
Acronym: TOBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cantonal Hospital, Frauenfeld (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Volker Viereck, Prof. Dr., Cantonal Hospital, Frauenfeld
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOL-OAB-01-08
Record Dates: First submitted 2011-01-21; First posted 2011-03-15 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; urinary frequency
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- solifenacin 5mg, PFMT and WBVT (Experimental): Patients randomized to group A will receive solifenacin 5mg tablet once daily and a training programme for PFMT and WBVT once a week.
  Interventions: Drug: solifenacin; Procedure: PFMT and WBVT
- solifenacin 5mg (Active Comparator): Subjects randomised to group B will receive solifenacin 5mg tablet once daily.
  Interventions: Drug: solifenacin

INTERVENTIONS:
Drug: solifenacin — solifenacin 5mg tablet once daily
  Other Names: brand name: vesicare
Procedure: PFMT and WBVT — pelvic floor muscle and whole body vibration training once a week
  Other Names: Pelvic Floor Muscle Training; Whole Body Vibration Training; Galileo
  Arms: solifenacin 5mg, PFMT and WBVT

SUMMARY:
The aim of the present study is to investigate in patients with overactive bladder syndrome (OABS) whether a combination treatment of solifenacin with pelvic floor muscle training and whole body vibration training achieves a better treatment outcome than a treatment with solifenacin alone.

DETAILED DESCRIPTION:
The treatment of patients with OAB in clinical practice often consists of drug therapy in combination with bladder training and/or behavioural therapies such as whole body vibration training (WBVT) and pelvic floor muscle training (PFMT). However, very little data exist on the benefits of such combinations. In particular, there are not data on the association of antimuscarinic agents with both WBVT and PFMT. In order to optimize the treatment of OAB it is of great importance to conduct studies which compare pharmacotherapy alone with a combination of pharmacotherapy and behavioural techniques.

The aim of the present study is to investigate in patients with OABS whether a combination treatment of solifenacin with pelvic floor muscle training and whole body vibration training achieves a better treatment outcome than a treatment with solifenacin alone.

At the baseline visit subjects will be randomised into 2 treatment arms. Patients randomized to group A will receive solifenacin 5mg tablet once daily and a training programme for PFMT and WBVT once a week. Subjects randomised to group B will receive solifenacin 5mg tablet once daily. Efficacy evaluation will take place at week 8 and 16. Safety evaluations will take place at each visit. At week 8, after discussion with the investigator, the patient will have an option to continue with the original dose or request a dose increase based on their satisfaction of efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with symptoms of overactive bladder (urinary frequency and urgency with or without incontinence) for ≥ 3 months
* Age ≥ 18 years old
* Urinary frequency ≥ 8 micturitions on average per 24 hours during the 3-day micturition diary period
* At least 3 episodes of urgency with or without incontinence (≥ 3) during the 3-day micturition diary period
* Patient provides written informed consent
* Patient is willing to complete the micturition diary

Exclusion Criteria:

* Clinically significant bladder outflow obstruction at risk of urinary retention (at the discretion of the investigator)
* Significant post void residual volume (> 200ml)
* Uncontrolled narrow angle glaucoma, urinary or gastric retention, severe ulcerative colitis, toxic megacolon, myasthenia gravis or any other medical condition which in the opinion of the investigator makes the use of anticholinergics contraindicated
* Neurological cause of abnormal detrusor activity
* Any clinically significant condition, which in the opinion of the investigator makes the subject unsuitable for the study
* Current non-drug treatment including pelvic floor muscle and whole body vibration training
* Known contraindications for whole body vibration training (cardiovascular, neurological or orthopaedic diseases, diabetes, tumor, pacemaker)
* Pregnant women or women who intend to become pregnant during the study
* Known or suspected hypersensitivity to solifenacin or lactose
* Concomitant use of a strong cytochrome P450 3A4 inhibitor (e.g. ketoconazole)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change of patient perception of bladder condition (PPBC) | baseline and 16 weeks
  The primary efficacy parameter is the change from baseline in mean score of patient perception of bladder condition (PPBC). Between-treatment differences in changes from baseline to endpoint will formally be tested using an analysis of variance (ANOVA).
  For the primary efficacy parameter, statistically significant superiority of solifenacin combined with pelvic floor muscle training (PFMT) and whole body vibration training (WBVT) to solifenacin alone must be obtained.

SECONDARY OUTCOMES:
Change in micturitions/24h based on a 3-day micturition diary | baseline and 16 weeks
  The analysis as described for the primary endpoint will be also applied for the secondary variables:
  Change from baseline in mean score of number of micturitions/24h based on a 3-day micturition diary.
Change of urgency episodes (grade ≥3) /24h | baseline and 16 weeks
  The analysis as described for the primary endpoint will be also applied for the secondary variables:
  Change from baseline in mean number of urgency episodes (grade ≥3) /24h.
Change in volume voided per micturition | baseline and 16 weeks
  The analysis as described for the primary endpoint will be also applied for the secondary variables:
  Change from baseline in mean volume voided per micturition.
Change in number of incontinence and urge incontinence episodes/24h | baseline and 16 weeks
  The analysis as described for the primary endpoint will be also applied for the secondary variables:
  Change from baseline in mean number of incontinence and urge incontinence episodes/24h.
Change in number of pads used/24h | baseline and 16 weeks
  The analysis as described for the primary endpoint will be also applied for the secondary variables:
  Change from baseline in mean number of pads used/24h.

CONTACTS AND LOCATIONS:
Overall Officials: Volker VV Viereck, physican, Principal Investigator — Cantonal Hospital, Frauenfeld
Locations (1):
- Blasenzentrum, Cantonal Hospital, Frauenfeld, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: No